CLINICAL TRIAL: NCT05861271
Title: Adjuvant Pyrotinib and Capecitabine For HER2 Positive Micro Invasive Breast Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhimin Shao, Director of General Surgery of Fudan Shanghai Cancer Center, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HERMIONE
Record Dates: First submitted 2023-05-07; First posted 2023-05-16 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Breast Cancer Stage I
MeSH Terms: conditions — Breast Neoplasms | interventions — pyrotinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm-1 (Experimental): Pyrotinib: 400mg QD Po for half a year, and Capecitabine: 500mg Tid Po for half a year Use of endocrine drugs in endocrine receptor (HR)-positive patients after chemotherapy. For premenopausal patients: tamoxifen (10 mg po, bid, for 5 years) or toremifene (60 mg po, qd, for 5 years); for postmenopausal patients: letrozole (2.5 mg, po, qd for 5 years) or anastrozole (1 mg, po, qd for 5 years) or exemestane (25 mg, po, qd for 5 years).
  After chemotherapy, radiation therapy will be started if necessary.
  Interventions: Drug: Capecitabine，Pyrotinib
- Arm-2 (No Intervention): No adjuvant chemotherapy or targeted therapy. Use of endocrine drugs in endocrine receptor (HR)-positive patients after chemotherapy. For premenopausal patients: tamoxifen (10 mg po, bid, for 5 years) or toremifene (60 mg po, qd, for 5 years); for postmenopausal patients: letrozole (2.5 mg, po, qd for 5 years) or anastrozole (1 mg, po, qd for 5 years) or exemestane (25 mg, po, qd for 5 years).
  After chemotherapy, radiation therapy will be started if necessary.

INTERVENTIONS:
Drug: Capecitabine，Pyrotinib — Pyrotinib and Capecitabine for half a year
  Other Names: Pyrotinib
  Arms: Arm-1

SUMMARY:
For patients with HER2-positive early-stage breast cancer, NCCN guidelines recommend chemotherapy plus targeted therapy as the standard adjuvant treatment for patients with tumors larger than 1 cm or lymph node-positive. The APT study enrolled patients with stage I HER2-positive breast cancer and has confirmed the efficacy and safety of intravenous chemotherapy combined with targeted therapy, but only 2.2% of the patients enrolled in microinvasion are enrolled, and there is a lack of large sample size data to provide a treatment reference for these patients. In order to further explore the optimal strategy for adjuvant therapy in this type of patient, we designed a new clinical trial to evaluate the efficacy and safety of oral capecitabine plus pyrotinib as adjuvant therapy in previous retrospective studies.

ELIGIBILITY:
Inclusion Criteria:

1. Women aged 18-70;
2. The pathology of early breast cancer after surgery is T1micN0: histologically confirmed that the longest diameter of invasive cancer does not exceed 1mm or the maximum diameter of multiple invasive lesions is less than 1mm, and the lymph node is negative (N0);
3. The pathological type of immunohistochemistry needs to meet the following conditions: HER-2 (3+) or HER-2 (0-2+) but amplified by FISH detection.
4. Hormone receptor negative (HR-) is defined as ER, PR expression is <1%; Hormone receptor positivity (HR+) is defined as ER and/or PR expression ≥1%.
5. For patients with both invasive lesions, if both lesions are HER-2 positive, they can be enrolled.
6. ECOG score≦ 1 point;
7. No obvious dysfunction of major organs;
8. Blood routine: ANC ≥1.5×109/L, PLT≥100×109/L, blood Hb≥ 9 g/dl (no transfusion within 14 days);
9. Liver function: total bilirubin ≤1.25×ULN; AST and ALT <2.5×ULN;
10. Renal function: creatinine clearance ≥ 50 mL/min, blood creatinine ≤ 1.5 ×ULN;
11. Cardiac function: ECG is generally normal, QTc< 470 ms; LVEF > 50%;
12. contraception during treatment for women of childbearing age;
13. No history of other malignant tumors in the past 5 years;
14. With the consent of the person and signed the informed consent form, or signed by the patient's legal representative with the authorization of the patient.
15. Can be followed up and good compliance.

Exclusion Criteria:

1. The maximum size of the infiltrate is more than 1mm in diameter or the axillary lymph node is positive
2. HER2 negative: immunohistochemical HER2-,+; Immunohistochemical HER2+ while FISH has no amplification;
3. Patients who have received neoadjuvant therapy or any other form of systemic therapy or local therapy other than surgery, including chemotherapy, targeted, radiotherapy, or endocrine therapy, prior to enrollment
4. History of other malignant tumors, except cured basal cell carcinoma of the skin and carcinoma in situ of the cervix;
5. Metastasis of any part;
6. Pregnant or lactating women, women of childbearing age who cannot be effectively contraceptives;
7. Patients who participate in other clinical trials at the same time;
8. Severe organ function (heart, lung, liver and kidney) insufficiency, LEVF < 50% (ultracardiogram); severe cardiovascular and cerebrovascular diseases (such as: unstable angina, chronic heart failure, uncontrollable hypertension >150/90mmgh, myocardial infarction or cerebrovascular accident) within 6 months before enrollment; diabetics with poor glycemic control; Patients with severe hypertension;
9. Severe or uncontrolled infection;
10. Those who have a history of psychotropic substance abuse and cannot quit or have a history of mental disorders;
11. Patients who are judged by the investigator to be unsuitable to participate in this study.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1008 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
iDFS | 5 years
  invasive disease-free survival

SECONDARY OUTCOMES:
DDFS | 5 years
  distant disease free survival
OS | 5 years
  overall survival

CONTACTS AND LOCATIONS:
Locations (1):
- Breast cancer institute of Fudan University Cancer Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided